CLINICAL TRIAL: NCT04215926
Title: The Epidemiological Investigation and Pathogenesis of NAFLD in HIV-infected Patients: a Cross-sectional Study
Brief Title: NAFLD in HIV-infected Patients
Acronym: NAFLDIH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Hongzhou Lu, professor, Shanghai Public Health Clinical Center
Other Study IDs: 20191126V2
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: HIV-infection/Aids; NAFLD
Keywords: HIV infection; NAFLD
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Non-alcoholic Fatty Liver Disease; HIV Infections | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and fecal sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-monoinfected outpatients: No intervention; cross-sectional study
  Interventions: Other: No intervention; cross-sectional study

INTERVENTIONS:
Other: No intervention; cross-sectional study — No intervention; cross-sectional study

SUMMARY:
The prevalence of NAFLD (nonalcoholic fatty liver disease) in HIV-infected patients is higher than that in general population, but the causes of morbidity and pathogenesis have not been fully explored. The investigators are planning to consecutively enroll 400 cases HIV-positive outpatients, and to detect NAFLD by ultrasound. The fecal and blood samples were also collected to explore the mechanism of NAFLD. The investigators aimed to determine the prevalence and risk factors of NAFLD in HIV infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~70 y;
* HIV-positive patients;
* written the informed consent

Exclusion Criteria:

* coinfected with HBV, HCV;
* secondary causes of fatty liver (eg, consumption of amiodarone and tamoxifen) and decompensated liver disease;
* significant alcohol consumption (>20 g per day for man, >10 g per day for woman);
* received antibiotics in preceding two months;
* autoimmune disease;
* severe heart, lung, kidney, brain, blood diseases or other important systemic diseases;
* pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected outpatients who was not coinfected with other form of viral hepatitis or drug induced liver disease, some severe systematic disease
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
morbidity of nonalcoholic fatty liver disease | 1 month
  NAFLD was diagnosed using ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu W, Liu D, Zhang R, Chen J, Shen Y. Prevalence and Risk Factors of Liver Fibrosis Among People With HIV and Metabolic Dysfunction-Associated Steatotic Liver Disease. Open Forum Infect Dis. 2025 Jul 2;12(7):ofaf369. doi: 10.1093/ofid/ofaf369. eCollection 2025 Jul. PMID 40667432